CLINICAL TRIAL: NCT02434484
Title: Post-Marketing Surveillance of Symbenda Injection (Bendamustine Hydrochloride) in Korean Patients
Brief Title: Symbenda Post-Marketing Surveillance (PMS)
Status: Completed | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: B0501-M065-501
Record Dates: First submitted 2015-04-28; First posted 2015-05-05 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphocytic Leukemia; Multiple Myeloma
Keywords: Symbenda; Non-Hodgkin's lymphomas; Chronic lymphocytic leukemia; Multiple myeloma; Bendamustine Hydrochloride
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphoid; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symbenda: Subjects who are prescribed with Symbenda per approved prescribing information of Symbenda will be enrolled in the study.

SUMMARY:
This is a PMS of Symbenda Injection (bendamustine hydrochloride) in Korean Patients. The main objective is to obtain safety information related to Symbenda treatment from clinical practice.

ELIGIBILITY:
Subjects who are prescribed with Symbenda per approved prescribing information of Symbenda will be enrolled in the study.

This study will be conducted as complete surveillance method; subjects who meet the inclusion/exclusion criteria and administrate Symbenda for the first time after conclusion of agreement will be enrolled.

Inclusion Criteria:

Patients who meet the following criteria will be eligible for inclusion in the study:

1. Patients with approved indication for Symbenda in Korea
2. Patients who have verbal or written consent for use of personal and medical information for the study purpose Investigators will refer to approved indications and contraindications regarding inclusion criteria.

Exclusion Criteria:

Investigators will refer to approved indications and contraindications regarding exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who are prescribed with Symbenda per approved prescribing information of Symbenda will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Safety of Symbenda as a measure of number of participants with adverse events/serious adverse events/adverse drug reactions | Up to 6 months
  An adverse event is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A serious adverse event is defined as any adverse event occurring at any dose that results in any of the following outcomes: results in death; is life threatening; results in inpatient hospitalization or prolongation of existing hospitalization; results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life function; results in a congenital anomaly/birth defect; or can be defined as any other important medical event.

SECONDARY OUTCOMES:
Non-Hodgkin's lymphomas response rate per Standardize Response Criteria for Non-Hodgkin's lymphomas to assess the tumor response | After 2nd cycle (each cycle = 28 days) up to 1.5 months
  Non-Hodgkin's lymphoma(NHL) is a cancer that starts in cells called lymphocytes, which are part of the body's immune system. Lymphocytes are in the lymph nodes and other lymphoid tissues (such as the spleen and bone marrow). Non-hodgkin's lymphoma is classified with two broad categories, such as high-grade or aggressive and low-grade or indolent.
  Response criteria for non-Hodgkin's lymphomas will be used to assess tumor response.
Chronic lymphocytic leukemia response rate per National Cancer Institute-Sponsored Working Group (NCISWG) criteria to assess the tumor response | After 2nd cycle (each cycle = 28 days) up to 2 months
  Chronic lymphocytic leukemia is a type of cancer that starts from cells that become lymphocytes in the bone marrow. The cancer (leukemia) cells start in the bone marrow but then migrate into the blood. NCISWG criteria will be used to assess tumor response.
Multiple myeloma response rate per International Myeloma Working Group (IMWG) uniform response criteria to assess the tumor response | After 2nd cycle (each cycle = 28 days) up to 2 months
  Multiple myeloma is a cancer formed by malignant plasma cells. Normal plasma cells are found in the bone marrow and are an important part of the immune system. IMWG Uniform Response Criteria will be used to assess tumor response.

CONTACTS AND LOCATIONS:
Locations (9):
- South Korea (9):
  - Eisai Trial Site #7, Busan
  - Eisai Trial Site #8, Busan
  - Eisai Trial Site #6, Daegu
  - Eisai Trial Site #4, Daejeon
  - Eisai Trial Site #5, Daejeon
  - Eisai Trial Site #9, Incheon
  - Eisai Trial Site #1, Seoul
  - Eisai Trial Site #2, Seoul
  - Eisai Trial Site #3, Seoul